CLINICAL TRIAL: NCT02511483
Title: Contribution of COMT Haplotypes in Propranolol Analgesic Efficacy for Treating Post-surgical Pain After Laparoscopic Hemicolectomy
Brief Title: Genetic Predictors of Analgesic Efficacy of Propranolol for Treating Postoperative Pain
Acronym: PRO_GENE_POP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Franco Carli, Professor of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-169-MUHC
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: COMT; Beta-blocker; Hemicolectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Propranolol; Analgesia, Patient-Controlled; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV-PCA morphine + Placebo PO (Placebo Comparator): Pain control after surgery will be performed through IV-PCA morphine. Placebo will be administered with the same schedule of Propranolol in the experimental arm.
  Parallel evaluation of Quantitative Sensory Testing (QST), Psychometric assessment and COMT-haplotypes will be included along the trial.
  Interventions: Drug: IV-PCA morphine; Drug: Placebo PO; Procedure: Quantitative Sensory Testing (QST); Other: Psychometric assessment; Genetic: COMT-haplotypes
- IV-PCA morphine + Propranolol PO (Experimental): The morning of the surgery a dose of Propranolol 20 mg PO will be administered. After surgery pain control will be performed with IV-PCA morphine; in addition a second dose of Propranolol 20 mg PO will be administered .
  During the first and second postoperative day Propranolol 30 mg PO (BID) will be administered. Parallel assessment of Quantitative Sensory Testing (QST), Psychometric assessment and COMT-haplotypes will be included along the trial.
  Interventions: Drug: Propranolol PO; Drug: IV-PCA morphine; Procedure: Quantitative Sensory Testing (QST); Other: Psychometric assessment; Genetic: COMT-haplotypes

INTERVENTIONS:
Drug: Propranolol PO — 20 mg PO BID Day of Surgery, 30 mg PO BID Day I and Day II post-op.
  Other Names: CAS No 525-66-6, DINs: 00740675, 00496480
  Arms: IV-PCA morphine + Propranolol PO
Drug: IV-PCA morphine — Morphine delivered via IV-PCA pump for 48 hours after surgery with standard program: bolus 1 mg, lock out 7 minutes, no background infusion.
  Other Names: Patient controlled Analgesia with intravenous morphine
Drug: Placebo PO — Placebo tablets administered with the same schedule of Propranolol tablets
  Other Names: tablet containing microcrystalline cellulose
  Arms: IV-PCA morphine + Placebo PO
Procedure: Quantitative Sensory Testing (QST) — Assessment of PPT (Pressure Pain Threshold) by pressure algometer and assessment of the post-op area of hyperalgesia by von Frey hair no. 16.
  Other Names: Pressure Pain Threshold and Hyperalgesia test
Other: Psychometric assessment — Questionnaires assessing for sleep quality (PSQI: Pittsburgh Sleep Quality Index), pain quality (sfMGPQ-Short Form-McGill Pain Questionnaire), somatization-depression-anxiety (SCL-90-R: Symptom Checklist 90 Revised), evolution of post-operative chronic pain (PQRS: Post-operative Quality of Recovery Scale)
  Other Names: PSQI, sfMGPQ, SCL-90-R, PQRS
Genetic: COMT-haplotypes — Assessing of High Pain Sensitivity (HPS), Average Pain Sensitivity (APS) and Low Pain Sensitivity (LPS) haplotypes for COMT by genotyping peripheral blood samples.
  Other Names: HPS, APS, LPS

SUMMARY:
This study is a randomized, double-blind, placebo controlled clinical trial. The main purpose of this study is to determine if postsurgical pain ratings are improved with treatment with oral Propranolol, and if the effectiveness of treatment can be modified by the presence or absence of SNPs (Single Nucleotide Polymorphism) associated with Cathecol-O-MethylTransferase (COMT) and mu-opioid receptor (MOR1) activity. The treatment period will last for three days and the observation period will last for six months. Effectiveness of treatment will be assessed by means of morphine consumption through quantitative evaluation of IV-PCA (Patient Controlled Analgesia) morphine as primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic hemicolectomy surgery.
* Self-reported Caucasians.
* ASA (American Society of Anesthesiologists) physical status of I or II.
* Agrees to provide signed and dated informed consent form.
* Willingness to agree with the Biobanking policy.

Exclusion Criteria:

* Uncontrolled medical or psychiatric conditions.
* Severe mental impairment.
* History of major depressive disorder, psychotic disorder or schizophrenia, and/or manic episodes within the past year.
* Active alcoholism within the past 6 months.
* Psychoactive recreational drug abuse within the past 6 months including MDMA, Ketamine, hallucinogens such as LSD and/or sympathomimetics such as Cocaine.
* Inability to comprehend pain assessment.
* Pregnancy and/or breast-feeding.
* Known hypersensitivity to Beta Blockers or Opioids.
* Currently taking Propranolol.
* Currently taking other hypotensive treatments.
* Currently taking Opioids.
* Patients with asthma or reactive airway disease.
* Patients with cardiac arrhythmia, coronary artery disease, congestive heart failure.
* Patients with renal failure or dialysis.
* Patients with liver insufficiency.
* Heart rate less than 60bpm or diastolic blood pressure <50 mmHg during the preoperative visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2016-11-12 (Actual)

PRIMARY OUTCOMES:
Total morphine delivered by IV-PCA | Day II Post-op

SECONDARY OUTCOMES:
Pressure Pain Threshold by digital pressure algometer | Pre-op visit, Day I Post-op, Day II Post-op, four weeks Post-op
Hyperalgesia test by von Frey hair | Pre-op visit, Day I Post-op, Day II Post-op, four weeks Post-op
Pain measured by the Numerical pain Rating Scale | Pre-op visit, one evaluation during the first 8 Post-op hours, Day I Post-op, Day II Post-op, 4 weeks Post-op, 3 month Post-op, 6 months Post-op
Somatization, depression and anxiety by SCL-90-R subscales | Pre-op visit
  Symptom Checklist 90 Revised (SCL-90-R) subscales for somatization, depression and anxiety
Sleep quality by PSQI | Pre-op visit, 4 weeks Post-op, 3 months Post-op, 6 months Post-op
  Pittsburgh Sleep Questionnaire Index (PSQI)
Pain quality by sfMGPQ | one evaluation during the first 8 Post-op hours, Day I Post-op, Day II Post-op
  Short Form-McGill Pain Questionnaire
Post-operative Chronic Pain by PQRS | Pre-op visit, Day II Post-op, 4 weeks Post-op, 3 months Post-op, 6 months Post-op
  Post-operative Quality of Recovery Scale (PQRS)

OTHER OUTCOMES:
COMT-haplotypes by blood sampling genotyping | Pre-op, Day III Post-op, 4 weeks Post-op

CONTACTS AND LOCATIONS:
Overall Officials: Luda Diatchenko, Professor, Principal Investigator — Anesthesia Department McGill University
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Background] Orrey DC, Halawa OI, Bortsov AV, Shupp JW, Jones SW, Haith LR, Hoskins JM, Jordan MH, Bangdiwala SI, Roane BR, Platts-Mills TF, Holmes JH, Hwang J, Cairns BA, McLean SA. Results of a pilot multicenter genotype-based randomized placebo-controlled trial of propranolol to reduce pain after major thermal burn injury. Clin J Pain. 2015 Jan;31(1):21-9. doi: 10.1097/AJP.0000000000000086. PMID 25084070
- [Background] Tchivileva IE, Lim PF, Smith SB, Slade GD, Diatchenko L, McLean SA, Maixner W. Effect of catechol-O-methyltransferase polymorphism on response to propranolol therapy in chronic musculoskeletal pain: a randomized, double-blind, placebo-controlled, crossover pilot study. Pharmacogenet Genomics. 2010 Apr;20(4):239-48. doi: 10.1097/FPC.0b013e328337f9ab. PMID 20216107
- [Background] Zaugg M, Tagliente T, Lucchinetti E, Jacobs E, Krol M, Bodian C, Reich DL, Silverstein JH. Beneficial effects from beta-adrenergic blockade in elderly patients undergoing noncardiac surgery. Anesthesiology. 1999 Dec;91(6):1674-86. doi: 10.1097/00000542-199912000-00020. PMID 10598610
- [Background] Schweinhardt P, Abulhasan YB, Koeva V, Balderi T, Kim DJ, Alhujairi M, Carli F. Effects of intravenous propranolol on heat pain sensitivity in healthy men. Eur J Pain. 2013 May;17(5):704-13. doi: 10.1002/j.1532-2149.2012.00231.x. Epub 2012 Oct 16. PMID 23070986
- [Background] Pranevicius M, Pranevicius O. Non-opioid anesthesia with esmolol avoids opioid-induced hyperalgesia and reduces fentanyl requirement after laparoscopy. Anesth Analg. 2009 Mar;108(3):1048. doi: 10.1213/ane.0b013e3181938f3f. No abstract available. PMID 19224829
- [Background] Chia YY, Chan MH, Ko NH, Liu K. Role of beta-blockade in anaesthesia and postoperative pain management after hysterectomy. Br J Anaesth. 2004 Dec;93(6):799-805. doi: 10.1093/bja/aeh268. Epub 2004 Sep 17. PMID 15377583
- [Background] Chen YW, Chu CC, Chen YC, Hung CH, Wang JJ. Propranolol elicits cutaneous analgesia against skin nociceptive stimuli in rats. Neurosci Lett. 2012 Aug 30;524(2):129-32. doi: 10.1016/j.neulet.2012.07.036. Epub 2012 Jul 26. PMID 22842397
- [Background] Zhang F, Tong J, Hu J, Zhang H, Ouyang W, Huang D, Tang Q, Liao Q. COMT gene haplotypes are closely associated with postoperative fentanyl dose in patients. Anesth Analg. 2015 Apr;120(4):933-40. doi: 10.1213/ANE.0000000000000563. PMID 25532715
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663